CLINICAL TRIAL: NCT06868329
Title: Effect of Using VR Game-based Training to Correct Lumbar Lordosis in Patients With Chronic Low Back Pain and Lumbar Hyperlordosis: Randomized Controlled Trial
Brief Title: Virtual Reality Vased Exercises and Hyperlordosis in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, Associate Professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2025-675
Record Dates: First submitted 2025-03-07; First posted 2025-03-10 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-03

CONDITIONS: Hyperlordosis
Keywords: lordosis; low back pain; lumbar curve; virtual reality; TBed
MeSH Terms: conditions — Swayback; Lordosis; Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All research-involved personnel will be concealed to the initial allocation of the patients to groups. The allocation process will be conducted by an administrative employer not involved in the assessment nor treatment. Permuted blocks method of randomization (block size 4 and 6) was used to ensure 1:1 allocation ratio. The numbers. Blinding will be assured by giving each participant a code number that will be used throughout the study. The therapist will only be allowed to reveal the interpretation of the code to allow him to provide the appropriate intervention. Patients, the assessor, and the statistician will be kept blind throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR TBed group (Experimental): this arm will receive superficial moist heat, hamstring and low back stretching plus posterior pelvic tilting exercises applied using TBed virtual reality gaming system,
  Interventions: Other: Superficial moist heat; Other: Hamstring and back muscles stretching; Other: Postural correction with lumbar stabilization using TBed
- Control group (Active Comparator): this arm will receive superficial moist heat, hamstring and low back stretching plus posterior pelvic tilting exercises applied using the traditional technique from supine position
  Interventions: Other: Superficial moist heat; Other: Hamstring and back muscles stretching; Other: posterior pelvic tilting exercises regular procedures

INTERVENTIONS:
Other: Superficial moist heat — Twenty minutes of automatic moist hot pack (Besmed© BE-267, Taiwan) of suitable size was used to apply superficial heat. The heat level was adjusted to the medium level. While the moist environment was assured by placing a moist sponge layer between the pack and its cotton outer coverage. The duration was calculated after 8 minutes of warming up (when the temperature reaches its maximum level). The patient-reported sensation should be moderate warmth. A thermal sensation test using two test tubes was performed before applying heat therapy to avoid any adverse effects
Other: Hamstring and back muscles stretching — Patients received manual passive stretch for the hamstring and lower back muscles. Three repetitions per session with every repetition sustained for 30 s. The patient assumed a long sitting position with both knees in full extension and feet together. The patient was then asked to bend forward from the hips to reach the furthest point towards the feet. The therapist applied over pressure by pressing hands on the patient's upper back and pushing forward.
Other: posterior pelvic tilting exercises regular procedures — Patients will be asked to assume the supine position with both knees semi-flexed. A small billow will be placed under the low back, another billow will be placed under the flexed knees for comfort. The patient will be asked to tuck the abdominal muscles inward and press with the low back on the underlying billow and hold for six seconds, then relax. after a few seconds of rest, the patient should repeat this procedure for 3 sets X 10 repetitions per session during the first 2 weeks. the number of sets will be increased according to the adaptation of each patient and his/her fatigue threshold.
  Arms: Control group
Other: Postural correction with lumbar stabilization using TBed — These exercises consisted of pelvic rocking, and activation of the upper back and interscapular muscles. TBed from Techno body©, Italy was used to assist the patient to perform these exercises through VR video gaming interface. The patients in the experimental group will be asked to contract the targeted muscles and push down on the surface of the TBed. Patient's pressure will activate the sensors inserted inside the TBed, which will be reflected on the game as triggering of the gun that targets flying fruits. The game consists of three levels, easy, medium, and hard. The patient will be asked to play the game for the lower back where pushing the lower back against the bed (posterior pelvic tilting) triggered the gun and for the upper back where pushing the scapula against the bed was the triggering action.
  Arms: VR TBed group

SUMMARY:
this study aimed to evaluate the impact of incorporating postural correction exercises through VR video gaming on lumbar lordotic angle (LLA), pain, range of motion (ROM), and function in patients with chronic non-specific low back pain (CNLBP). Furthermore, the study sought to assess satisfaction and commitment levels when VR was integrated into the exercise regimen

DETAILED DESCRIPTION:
Low back pain is referred to as the most common musculoskeletal dysfunction. Almost every person is at risk of experiencing a low back pain attack at least once in life. Due to its high prevalence rate, low back pain can be attributed to high rates of work absenteeism, long-term functional disability and compromised quality of life. A huge economic burden has been linked to the management of this condition, especially in low-income countries.

The mechanism of development of low back pain could be quite variable. Some cases develop low back pain after accidents or trauma to the lower spine or pelvis. In other occasions, bad postural alignment, such as anterior pelvic tilting, leg length discrepancy, could be the primary source of the lesion. Other patients could experience low back pain secondary to discogenic lesion in the lumbar spine, which is usually associated with referred pain to the lower extremities (sciatica). Interestingly, the majority of the cases have no obvious mechanism of origin. Hence, were referred to as nonspecific low back pain.

According to previous literature, some researchers argue that the lumbar spine lordotic curvature (LLC) is the origin of low back pain. This curve was developed in the early infancy when the infant starts to assume an upright posture. The presence of the LLC allows the center of mass of the trunk to be located superior to the hips and provides biomechanical advantages to the soft tissue in neutralizing shear loads and allows better locomotion on the lower extremity. However, this comes with the cost of increased susceptibility for the development of low back pain.

The value of the LLC is usually influenced by the surrounding muscles situated in the abdomen, low back, anterior and posterior hip region, and hamstrings. Imbalance between the sagittal plane muscles, such as tight low back muscle and anterior hip muscle along with weak or elongated abdominal muscles can result in anterior pelvic tilt and an increase in the LLC. Conversely, other patients might demonstrate a decrease in the LLC value secondary to muscle imbalance.

qLLC can be assessed accurately using plain X-ray of the spine. Several angles can be measured to reflect the LLC. However, the lumbar lordotic angle (LLA) is considered the most accurate one. LLA can be calculated using a lateral view X-ray film where the intersection angle between two lines was calculated. The first line was drawn from the upper surface of the first lumbar vertebra and the second line was drawn from the lower surface of the last lumbar vertebral body.

Due to the diverse mechanisms of low back pain, there are also variations of treatment strategies, exercise therapy, manual therapy, physical therapy modalities, as well as medications and surgery, which can be all used according to the characteristics of each patient.

Exercises consisting of pelvic rocking (anterior and posterior) are considered cornerstone in any exercise therapy because they improve mobility of the lower trunk muscles and regain balance between anterior and posterior muscle groups to regain the normal.

TBed is a fully sensorized treatment bed divided into four sections. It features a network of sensors capable of detecting any pressure applied by the patient's body, which is then displayed in real-time on an attached computer screen. This allows patients to play various games by using their neck, upper, and lower back muscles, making it an excellent option for video game-based rehabilitation of spinal conditions.

Numerous studies have explored the effectiveness of gaming and VR in treating low back pain (LBP), yet there remains debate about their short-term impact. Moreover, satisfaction and adherence to exercise sessions have not been thoroughly examined.

ELIGIBILITY:
Inclusion Criteria:

* males or females,
* 18 - 44 years of age,
* unilateral, bilateral, or central (midline) pain in the low back,
* demonstrate lumbar hyper lordosis of the lumbar spine (lumbar lordotic angle more than 40°, measured using flexi ruler and spinal mouse) (Tack 2021),
* pain persists for 3 months or more,
* pain intensity between 2 -6 on numeric pain rating scale (NPRS).

Exclusion Criteria:

* acute low back pain (less than 3 months),
* specific pain due to well diagnosed pathology such as trauma, surgery, dick lesion, tumor, adhesions.
* Low back pain associated with sciatica, patients who cannot stop using analgesic drugs during the period of the study.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Intensity of low back Pain | at base line and after 8 weeks of tretment
  Pain intensity will be assessed using NPRS. This scale consists of a horizontal 10cm line numbered from 0 to 10. The higher numbers indicate higher pain intensity while lower numbers indicate lower pain intensity. The validity and reliability of this scale for measuring musculoskeletal pain were approved in previous work. Participants were asked to select the number that represents their current pain level.
Active ROM of the lumbar spine | at base line and after 8 weeks of tretment
  Active Lumbar flexion and extension were assessed using the Back range of motion (BROM) device. This device was designed to assess the ROM of the lumbosacral region. It consisted of a set of inclinometers - attached to two plastic frames - arranged in vertical and horizontal fashions to assess the sagittal, frontal, and rotational movement of the lower back. BROM is a valid and reliable device for measuring lumbar ROM. The current study used BROM (Performance Attainment Associates, Roseville, Minnesota) to assess active flexion and extension of the lumbar spine. Measurements were taken according to the guidelines described previously.
  The AROM was determined by calculating the difference between the angle recorded in the starting position and the angle recorded at the end position of either flexion or extension.
Lumbar lordotic angle (LLA) | at base line and after 8 weeks of tretment
  LLA will be measured using a Flexi curve ruler. A flexi ruler is utilized as a non-invasive tool to assess lumbar curvature. This 60 cm ruler is constructed from special steel and coated with plastic, allowing it to be bent to match the lumbar curve and maintain its shape. Its reliability and validity have been previously confirmed. The assessment will be conducted by an assessor who will be unaware of the patient's intervention allocations. To measure the lumbar curve, patients will stand with their knees extended and feet about shoulder-width apart, while the lordosis was measured between the L1 and S2 prominences. The angle between L1 and S2, referred to as the Ө angle, will be calculated using the formula: Ө = 4[Arc tan (2H/L)], where L is the line connecting the two ends of the curve, and H is the maximum distance between L and the curve. The normal lordosis angle is 30 degrees, while angles exceeding 40 degrees are classified as hyper
Functional level | at base line and after 8 weeks of tretment
  The Oswestry Disability Index (ODI) was used to assess functional disability levels. It consists of 10 sections covering the discomfort of the back and the activities conducted every day. Each item has six answers with a score range from 0-5 according to the arrangement of the statement as 1st refers to 0 and the 2nd takes 1, etc. Then the scores were added to reach the total score ranging from 0 - 50. This score can be used as raw data or it can be used to calculate a percentage. In either case, lower values indicate better function and higher values indicate more disability. In the current study, the raw data was used to conduct the analysis, as it was considered more sensitive to show minor changes compared to ratio values. The validity and reliability of the ODI have been studied and shown to have a high level , where the ICC for the reliability range (0.96-0.88).

SECONDARY OUTCOMES:
Satisfaction level | after 8 weeks of tretment
  This outcome was measured using a 1-10 scale which resembles the NPRS. However, the 0 point indicated no satisfaction while the number 10 indicated maximum satisfaction. The patient was asked to answer the following question, "To what extent can you rate your satisfaction with the introduced physical therapy program?". The patient then chose any number from 0 to 10 that represented the current level of satisfaction
Commitment to exercise sessions | after 8 weeks of tretment
  This outcome was assessed by calculating the percentage (%) of the successful sessions that were attended by the patients and subdivided by 420 (the total number of sessions) and then multiplied by 100

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hail, Hail, Ha'il Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
data will be used in future studies